CLINICAL TRIAL: NCT03814473
Title: Eight Week ad Libitum Self-prepared Paleo Diet and Cardiometabolic Disease Risk Factors in Overweight Adults
Brief Title: Paleo Diet 8wk Feasibility in Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: Chatham University (Other)
Responsible Party: Principal Investigator, Melissa M Markofski, Asssitant Professor, University of Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000104
Record Dates: First submitted 2019-01-16; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary intervention (Experimental): All participants will follow an ad libitum self-administered Paleo diet for 8-weeks
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Participants provided with a brochure providing a thorough description of the diet, ~8 example recipes for each meal (i.e. breakfast, lunch, dinner, and snacks) included as a sample menu, and guidance to assist in shopping and self-preparation of food for the prescribed diet and to improve adherence. Diet consisted of following the popular "paleolithic" diet

SUMMARY:
Overweight, physically inactive but otherwise healthy adults habitually eating a traditional Western diet will follow an ad libitum self-administered Paleo diet for 8-weeks. Blood and body composition will be measured before and after the intervention period.

DETAILED DESCRIPTION:
The Paleo diet is a dietary method that is gaining popularity among the general population due to potential weight loss and disease prevention benefits. The feasibility of the Paleo diet and the effectiveness of self-administration in improving cardiometabolic disease risk factors remains uncertain. Examination od cardiometabolic disease risk factors in overweight, physically inactive adults before and after 8-weeks of an ad libitum self-administered Paleo dietary intervention. Methods: Overweight, physically inactive but otherwise healthy adults habitually eating a traditional Western diet follow an ad libitum self-administered Paleo diet for 8-weeks. Blood samples were analyzed for fasting cardiometabolic disease biomarkers. Participants complete three-day dietary recalls prior to, and during weeks 4 and 8 of the intervention to confirm Western diet consumption at pre-, track compliance, and to assess dietary changes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-55 years
* BMI > 25 kg/m2
* Currently consuming a typical Western diet (high carbohydrate, low fat diet), which will be assessed using the 3-day dietary record (public domain)

Exclusion Criteria:

* known cardiovascular, metabolic (including type I or type II diabetes), or respiratory disease
* smoking and/or smokeless tobacco users
* pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2015-04-14 (Actual); Study Completion 2015-04-14 (Actual)

PRIMARY OUTCOMES:
Serum cytokines | Change from pre-intervention (week zero) and post-intervention (upon completion of week 8)
  Serum measurement of interleukin (IL)-4 (pg/dL), IL-10 (pg/dL), interferon (INF)-gamma (pg/dL), tumor necrosis factor (TNF; pg/dL)
Serum growth factor | Change from pre-intervention (week zero) and post-intervention (upon completion of week 8)
  Serum measurement of brain derived neurotrophic factor (BDNF; ng/mL)
Serum biomarkers of energy homeostasis | Change from pre-intervention (week zero) and post-intervention (upon completion of week 8)
  Serum fibroblast growth factor (FGF)-21 (pg/mL) and adiponectin (pg/mL)
Serum glucose metabolism biomarkers | Change from pre-intervention (week zero) and post-intervention (upon completion of week 8)
  leptin (mg/dL), glucagon-like peptide (GLP)-1 (mg/dL), resistin (mg/dL), insulin (mg/dL), Gastric inhibitory polypeptide (GIP; mg/dL), glucagon (mg/dL), visfatin (mg/dL), ghrelin (mg/dL), plasminogen activator inhibitor (PAI)-1 (mg/dL), C-peptide (mg/dL)
Serum adipokines | Change from pre-intervention (week zero) and post-intervention (upon completion of week 8)
  Serum omentin (ng/mL) and nesfatin (ng/mL)

SECONDARY OUTCOMES:
Waist and hip circumference | Change from pre-intervention (week zero) and post-intervention (upon completion of week 8)
  Circumference of two midsection areas of the body (waist and hip) to estimate central adiposity
Subcutaneous body fat | Change from pre-intervention (week zero) and post-intervention (upon completion of week 8)
  Skin fold thickness (mm) of body fat
Dietary composition | Change from pre-intervention (week zero) and post-intervention (upon completion of week 8)
  3-day food diary to approximate macronutrient composition (grams)
Dietary energy intake | Change from pre-intervention (week zero) and post-intervention (upon completion of week 8)
  3-day food diary to approximate total energy intake (kcal)
Blood pressure | Change from pre-intervention (week zero) and post-intervention (upon completion of week 8)
  Measurement of blood pressure from the arm (mmHg)
Body weight | Change from pre-intervention (week zero) and post-intervention (upon completion of week 8)
  Measurement of participant's body weight (kg)
Body height | pre-intervention (week zero)
  Measurement of participant's height (m) to (along with body weight) calculate body mass index (kg/m^2)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Carrillo, Study Director — Chatham University
Locations (2):
- United States (2):
  - Chatham University, Pittsburgh, Pennsylvania
  - University of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
non-identifiable study variables (i.e. serum biomarkers) may be deposited in sharing databases for open access publications